CLINICAL TRIAL: NCT05832190
Title: Correcting GUT MicrobioTa by Combined Supplementation of FibERs and BIotiN to Improve Microbiome and Optimize Bariatric Surgery Outcomes
Acronym: GUTERRING
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: end of ERC funding period
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP220972; 2022-A02251-42 (Other: IDRCB)
Record Dates: First submitted 2023-02-10; First posted 2023-04-27 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Severe Obesity; Metabolic Syndrome
Keywords: GUT microbioTa; Supplementation; Fibers; Biotin; Microbiome; Bariatric surgery
MeSH Terms: conditions — Obesity, Morbid; Metabolic Syndrome | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1: patient with usual follow-up (standard of care) (Active Comparator): receiving during 3 months before the surgery usual general dietary recommendations regarding balanced diet comprising legumes and fruits, meat or equivalent, dairy products and starch and bread
  Interventions: Other: Standard of care
- Arm 2: Same usual general dietary recommendations PLUS Biotin (Experimental): Patients will receive the same usual general dietary recommendations PLUS 1 capsule per day of Biotin 450 µg per day during 3 months before the surgery.
  Interventions: Other: Standard of care; Dietary Supplement: Biotin supplement
- Arm 3: Same usual general dietary recommendations PLUS Fiber (Experimental): Patients will receive the same usual general dietary recommendations PLUS 3 servings per day of PureLean® Fiber, a powdered blend of fibers and prebiotics, during 3 months before the surgery
  Interventions: Other: Standard of care; Dietary Supplement: Fiber supplement
- Arm 4: Same usual general dietary recommendations PLUS Fiber PLUS Biotin (Experimental): Patients will receive the same usual general dietary recommendations PLUS 3 servings per day of PureLean® Fiber and Biotin 450 µg per day (1 capsule per day), during 3 months before the surgery.
  Interventions: Other: Standard of care; Dietary Supplement: Biotin supplement; Dietary Supplement: Fiber supplement

INTERVENTIONS:
Other: Standard of care — Patients receiving during 3 months before the surgery usual general dietary recommendations regarding balanced diet comprising legumes and fruits, meat or equivalent, dairy products and starch and bread
Dietary Supplement: Biotin supplement — 1 capsule per day of Biotin 450µg during 3 months before the surgery.
  Arms: Arm 2: Same usual general dietary recommendations PLUS Biotin; Arm 4: Same usual general dietary recommendations PLUS Fiber PLUS Biotin
Dietary Supplement: Fiber supplement — 3 servings per day of PureLean® Fiber, a powdered blend of fibers and prebiotics, during 3 months before the surgery
  Arms: Arm 3: Same usual general dietary recommendations PLUS Fiber; Arm 4: Same usual general dietary recommendations PLUS Fiber PLUS Biotin

SUMMARY:
Bariatric surgery improves health outcomes with a maximal weight loss on average occurring 1 year after surgery but with dramatic between-subjects variability in weight loss (ranging from 20 to 160% excess weight loss) for reasons that remain to be elucidated.

The investigators hypothesize that targeting the 3 months pre-surgery period by a calibrated dietary intervention, with fiber enrichment and biotin, will improve gut microbiota richness and subsequently improve subjects' metabolic health that may optimize post bariatric surgery outcomes.

The study is designed as a pilot, comparative, randomized, open-label trial with 4 arms: standard of care, biotin only, fibers only, biotin + fibers.

DETAILED DESCRIPTION:
This is a pilot open label study that aims to examine the efficacy of biotin supplementation with or without enriched soluble and insoluble fibers given during 3 months before the bariatric surgery, on gut microbiota composition and functional capacity to produce B vitamins (primary outcomes), compared to standard of care (e.g. patient preparation to bariatric surgery).

The study is a 4-arm clinical trial:

Arm 1: patients with usual follow-up (standard of care) receiving during 3 months before the surgery usual general dietary recommendations regarding balanced diet comprising legumes and fruits, meat or equivalent, dairy products and starch and bread Arm 2: Same usual general dietary recommendations PLUS Biotin 450 µg per day (1 capsule per day) during 3 months before the surgery.

Arm 3: Same usual general dietary recommendations PLUS 3 servings per day of PureLean® Fiber, a powdered blend of fibers and prebiotics, during 3 months before the surgery Arm 4: Same usual general dietary recommendations PLUS 3 servings per day of PureLean® Fiber and Biotin 450 µg per day (1 capsule per day), during 3 months before the surgery.

There will be two periods: period 1 during the 3 months before bariatric surgery and period 3 after bariatric surgery (usual standard of care follow-up). The 4 groups will be compared before bariatric surgery and up to 6 months afterward

Patients will receive a schedule of hospitalizations and visits before and after the surgery:

* V0: 3 months before surgery
* V1: presurgery visit, one day hospitalization
* V2: 3 months post-surgery
* V3: 6 months post-surgery
* V4:12 months post-surgery

At each visit (V0, V1, V2 , V3 and V4), will be performed as part of research:

* Adipose tissue aspiration
* Questionnaires
* Fecal samples
* Saliva samples (oral microbiota)
* Blood samples
* Urine samples This planning is part of the standard of care. The same follow-up will be performed in the 4 arms.

Patients will be called 3 times between V0 and V1 by dietician as part of research.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and < 60 years
2. BMI ≥ 40 kg/m² or BMI > 35 kg/m² with at least one comorbidity belonging to metabolic syndrome (hyperglycemia (fasting glycemia > 1g/l, Non diabetic with HbA1C<7% without antidiabetic treatment), dyslipidemia (HDL-cholesterol <0.5 g/l or receiving treatment against dyslipidemia), or increased blood pressure (SBP >13, DBP>9 or treated by antihypertensive drug)), or sleep apnoea, weight stable (less than 3 kg variation in the 2 months before
3. Usual Fiber intake < 20g/day in food consumption evaluated by 24h recall
4. Signature of the informed consent
5. Effective contraception in women of childbearing age
6. Subject with health insurance (except AME)

Exclusion Criteria:

1. Patients receiving antibiotics (ATB) at the selection time or within the 2 previous months.

   (if agreeing to participate to the study, the patients will be proposed randomization 3 months after stopping ATB)
2. Type 1 or type 2 diabetes
3. HIV, HBV, HCV
4. Gastrointestinal disease: Acute or chronic diarrhea (i.e. more than 3 liquid or fluid stools/day)
5. Previous history of gastrointestinal neoplasia or polyps
6. Factors that may affect the composition of the intestinal microbiota: Special Diet (exclusion diet, vegetarian diet), taking immunosuppressants (eg calcineurin inhibitors, corticosteroids, biological agents, etc.), taking transit modulators (osmotic or prebiotics such as lactulose).
7. Pregnancy or breastfeeding women
8. Subject under guardianship or curatorship
9. Subject deprived of their liberty by a judicial or administrative decision
10. Patient participating to another interventional clinical research (Jardé 1)
11. Subject physically unable to give his or her written consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2024-12-24 (Actual); Study Completion 2024-12-24 (Actual)

PRIMARY OUTCOMES:
3-month variation of gut microbiota richness 3 months after the start of the different dietary interventions | At the inclusion and 3 months after supplementation
  Access to gut microbiota richness will be provided after gut microbiota sequencing (by INRAE) with the acquisition of a table comprising the number of genes as well as the record of bacterial genes implicated in synthesis and transport of biotin. Based on preclinical observation, it is expected that the arm 4 combining biotin and fibers will show the highest richness

SECONDARY OUTCOMES:
Assess changes in body weight between the visit 3 months before surgery and the pre-surgery visit, the visit at 3 and 6 months after surgery. | At the inclusion, 3months after supplementation, 3, 6 and 12 months after surgery
  Body Weight will be obtained at each visit between 8 and 10 am using standardized procedures: Body weight will be obtained with a scale (Seca GmbH & Co., Hamburg, Germany) in kilograms
Assess changes in BMI between the visit 3 months before surgery and the pre-surgery visit, the visit at 3 and 6 months after surgery | At the inclusion, 3months after supplementation, 3, 6 and 12 months after surgery
  Height will be obtained with measuring scale rounded to the nearest 0.5 cm in centimeters Weight and height will be combined to report BMI in kg/m^2
Assess changes in waist circumference between the visit 3 months before surgery and the pre-surgery visit, the visit at 3 and 6 months after surgery | At the inclusion, 3 months after supplementation, 3, 6 and 12 months after surgery
  Twaist circumference will be measured in centimeters at the level of the iliac crest and hip circumference at the level of the symphysis-great trochanter to the nearest 1 cm.
Assess changes in fat mass between the visit 3 months before surgery and the pre-surgery visit, the visit at 3 and 6 months after surgery | At the inclusion, 3 month after supplementation, 3, 6 and 12 months after surgery
  For the measurement of fat mass (in kilograms and percentage of body weight), patients will undergo DEXA analysis, using the Hologic Inc. machine, QDR 4500W t using standard software (Hologic Inc., S/N 47168 VER. 11.2)
Assess changes in lean mass between the visit 3 months before surgery and the pre-surgery visit, the visit at 3 and 6 months after surgery | At the inclusion, 3 month after supplementation, 3, 6 and 12 months after surgery
  For the measurement of lean mass (in kilograms and percentage of body weight), patients will undergo DEXA analysis, using the Hologic Inc. machine, QDR 4500W t using standard software (Hologic Inc., S/N 47168 VER. 11.2)
Assess changes in visceral adipose tissue mass between the visit 3 months before surgery and the pre-surgery visit, the visit at 3 and 6 months after surgery | At the inclusion, 3 month after supplementation, 3, 6 and 12 months after surgery
  For the measurement of visceral adipose tissue mass (in kilograms and percentage of body weight), patients will undergo DEXA analysis, using the Hologic Inc. machine, QDR 4500W t using standard software (Hologic Inc., S/N 47168 VER. 11.2)
Assess changes in blood pressure between the visit 3 months before surgery and the pre-surgery visit, the visit at 3 and 6 months after surgery. | At the inclusion, 3 months after supplementation, 3, 6 and 12 months after surgery
  Blood pressure (Systolic and Diastolic) will be measured three times with a mercury sphygmomanometer in the right arm, with patients in a sitting position after five minutes of rest. The average of the three measurements will be considered for analysis
Assess changes in insulin resistance markers between the visit 3 months before surgery and the pre-surgery visit, the visit at 3 and 6 months after surgery. | At the inclusion, 3 months after supplementation, 3, 6 and 12 months after surgery
  To predict insulin resistance, homeostatic model assessment of insulin resistance (HOMA-IR) will be calculated according to the following formula: HOMA-IR = [fasting insulin (mU/l) x fasting blood glucose (mmol/l)]/22.5.
Assess changes in insulin sensitivity markers between the visit 3 months before surgery and the pre-surgery visit, the visit at 3 and 6 months after surgery | At the inclusion, 3 months after supplementation, 3, 6 and 12 months after surgery
  Quantitative insulin sensitivity check index (QUICKI) will be calculated according to the following formula: QUICKI= 1/[log(fasting insulin) + log(fasting blood glucose)
Assess change in Leptin between the visit 3 months before surgery and the pre-surgery visit, the visit at 3 and 6 months after surgery. | At the inclusion, 3 months after supplementation, 3, 6 and 12 months after surgery
  Leptin (ng/mL) will be measured according to standard protocols using human Leptin ELISA Kit (MyBioSource, Cod. MBS9425103)
Assess change in Adiponectin between the visit 3 months before surgery and the pre-surgery visit, the visit at 3 and 6 months after surgery. | At the inclusion, 3 months after supplementation, 3, 6 and 12 months after surgery
  Adiponectin (µg/mL) will be measured according to standard protocols using human Adiponectin /Acrp30 Quantikine ELISA kit (DRP300, R&D Systems)
Assess changes in glucose between the visit 3 months before surgery and the pre-surgery visit, the visit at 3 and 6 months after surgery | At the inclusion, 3 months after supplementation, 3, 6 and 12 months after surgery
  A fasting venous blood draw will be taken from a vein on the forearm to verify blood glucose (g/L) using commercial kits
Assess changes in lipid profile between the visit 3 months before surgery and the pre-surgery visit, the visit at 3 and 6 months after surgery | At the inclusion, 3months after supplementation, 3, 6 and 12 months after surgery
  A fasting venous blood draw will be taken from a vein on the forearm to verify triglycerides ( g/L), total cholesterol (g/L), HDL- cholesterol(g/L), LDL- cholesterol (g/L), using commercial kits
Assess changes in liver function between the visit 3 months before surgery and the pre-surgery visit, the visit at 3 and 6 months after surgery | At the inclusion, 3 months after supplementation, 3, 6 and 12 months after surgery
  A fasting venous blood draw will be taken from a vein on the forearm to verify alanine aminotransferase (ALT) (UI/L), aspartate aminotransferase (AST) (UI/L), gamma-glutamyl transferase (GGT) (UI/L), using commercial kits
Assess change in inflammatory marker (C-reactive protein) between the visit 3 months before surgery and the pre-surgery visit, the visit at 3 and 6 months after surgery. | At the inclusion, 3 months after supplementation, 3, 6 and 12 months after surgery
  C-reactive protein (mg/l) will be measured by multiplex analysis
Assess changes in inflammatory markers (IL6, sCD14, IL1b, IL10, TNF-R) between the visit 3 months before surgery and the pre-surgery visit, the visit at 3 and 6 months after surgery. | At the inclusion, 3 months after supplementation, 3, 6 and 12 months after surgery
  IL6, sCD14, IL1b, IL10, TNF-R (pg/mL) will be measured by multiplex analysis
Assess changes in adipose tissue gene expression for biotin-dependent carboxylases and inflammatory genes | At the inclusion, 3 months after supplementation, 3, 6 and 12 months after surgery
  Adipose tissue aspiration (100 mg): measure for adipose cell size and gene expression study (5-carboxylase depending of biotin and inflammatory markers).
Assess changes in quality of life | At the inclusion, 3 months after supplementation, 3, 6 and 12 months after surgery
  Information regarding their usual lifestyle by autoquestionnaire: SF-36 (Medical Outcome Study Short Form - 36) ranging from 0 to 100. A low score reflects a perception of poor health, loss of function, presence of pain. A high score reflects a perception of good health, an absence of functional deficit and pain
Assess changes in emotional eating | At the inclusion, 3 months after supplementation, 3, 6 and 12 months after surgery
  Information regarding their usual lifestyle by autoquestionnaire : Dutch Eating Behaviour Questionaire ( DEBQ) : this questionnaire is composed by 33 items divided into 3 scores. Of the original 100 items, 33 will be maintained and divided into 3 scores. Each question allows for 5 possible answers rated from 0 to 5 points. The possible answers are: never (1 point), rarely (2 points), sometimes (3 points), often (4 points), very often (5 points). The scores are as follows:
  * Restriction score: 10 questions on the "organised" will to control one's weight.
  * Emotionality score: 13 questions divided into two sub-scores, diffuse emotionality for 4 questions and definite emotionality for 9 questions
  * Externality score: 10 questions For each score, if the average of the responses is higher than 30, the subject is considered respectively: restricted, emotional eating or external.
Assess changes in physical activity | At the inclusion, 3 months after supplementation, 3, 6 and 12 months after surgery
  Information regarding their usual lifestyle by autoquestionnaire : Recent Physical Activity Questionnaire ( RPAQ) :
  * Interpretation of the physical activity (PA) level : Total sum week + weekend :
  * <8.3 MET.h/week: inactive ;
  * From 8.3 MET.h/week: active, with the possibility of two levels:
    * From 8.3 to 16.7: moderate PA;
    * >16.7: high PA.
  * interpretation of the time spent inactive : For weekdays and weekends:
  * ≤7h/d: non-sedentary ;
  * >7h/d: sedentary.
Assess changes in anxiety | At the inclusion, 3 months after supplementation, 3, 6 and 12 months after surgery
  Information regarding their usual lifestyle by autoquestionnaire : HAD questionnaire (Hospital Anxiety and Depression questionnaire) : the HAD scale is an instrument to screen for anxiety and depressive disorders. It consists of 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D). (total D), thus allowing two scores to be obtained (maximum score for each score = 21).
  For each of the scores (A and D):
  * 7 or less: no symptomatology
  * 8 to 10: doubtful symptomatology
  * 11 and more: definite symptomatology.
Assess changes in sleep quality | At the inclusion, 3 months after supplementation, 3, 6 and 12 months after surgery
  Information regarding their usual lifestyle by autoquestionnaire : STOP band (Snoring - Tired - Observed apnea - Pressure - BMI - Age - Neck size - Gender) questionnaire:
  Interpretation of the STOP-BANG:
  The STOP-BANG score can be used to identify subjects at risk of sleep apnea (S.A.).
  * Low risk of S.A.: Score from 0 to 2.
  * Moderate risk of S.A.: Score of 3 to 4.
  * High risk of S.A.: Score of 5 to 8, or STOP ≥ 2 and male sex, or STOP ≥ 2 and BMI > 35, or STOP ≥ 2 and neck circumference > 40cm.
Assess changes in stool consistency | At the inclusion, 3 months after supplementation, 3, 6 and 12 months after surgery
  Patients will be asked to answer a Bristol stool scale : the Bristol Scale has seven types of profiles, ranging from constipation (type 1 and 2) to diarrhea (type 6 and 7). Each type corresponds to a specific description of the stool.
Assess changes in stool inflammatory markers | At the inclusion, 3 months after supplementation, 3, 6 and 12 months after surgery
  Fecal calprotectin (in µg/g of feces) will be measured through ELISA kit
Change in gut microbiota composition by quantitative metagenomics. | At the inclusion, 3 months after supplementation, 3, 6 and 12 months after surgery
  Total fecal DNA will be extracted, sequenced by oxford nanopores technology and analysed using momr R package.
Change in intestinal permeability by Zonuline dosage | At the inclusion, 3 months after supplementation, 3, 6 and 12 months after surgery
  Zonuline dosage (ng/mL)
Change in intestinal permeability by LPS-binding protein dosage | At the inclusion, 3 months after supplementation, 3, 6 and 12 months after surgery
  LPS-binding protein dosage (mg/L)
Systemic measurement of Biotin (B8),B6 and B9-vitamins | At the inclusion, 3 months after supplementation, 3, 6 and 12 months after surgery
  Biotin (B8),B6 and B9 (nmol/L) will be measured by Elisa dosage from blood samples
Systemic measurement of B12-vitamin | At the inclusion, 3 months after supplementation, 3, 6 and 12 months after surgery
  B12 (pmol/L) will be measured by Elisa dosage from blood samples

CONTACTS AND LOCATIONS:
Locations (1):
- hôpital Pitié Salpêtrière, Paris, France, France

IPD SHARING:
Plan to Share IPD: No